CLINICAL TRIAL: NCT06426446
Title: Monitoring Patients With Severe Obesity Treated With Wegovy® Using Connected Device: Real-world Data
Acronym: TELE-SEMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: BPIfrance (Other); Withings (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP230587
Record Dates: First submitted 2024-05-13; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Obesity
Keywords: Obesity; Wegovy; Semaglutide 2.4 mg/week
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connected scale (Experimental): Patients receiving connected scale
  Interventions: Device: Withings Body Comp Pro

INTERVENTIONS:
Device: Withings Body Comp Pro — Withings Body Comp Pro from which the following features will be used: body weight, body composition (fat, muscle and bone mass, cardiovascular health (pulse wave velocity, arterial stiffness, vascular age, standing heart rate), nervous health (electrochemical skin conductance)

SUMMARY:
This study involves collecting real-world data on body weight, body composition, cardiovascular parameters, and neurovegetative parameters using a connected scale in patients with severe obesity treated with Wegovy®.

DETAILED DESCRIPTION:
Obesity is a chronic disease associated with numerous co-morbidities. New treatments for obesity, notably GLP-1 (Glucagon-like peptide 1) analogs, have led to promising advances. Semaglutide 2.4 mg weekly subcutaneous injection, marketed under the brand name Wegovy®, was recently approved in France for weight loss in patients with severe obesity and at least one comorbidity. Several real-world studies have confirmed the effectiveness of semaglutide in reducing body weight and HbA1c. However, few studies have evaluated the kinetics and interindividual variability of changes in body weight and composition as well as cardiovascular health. There appears to be a need for a comprehensive real-world assessment of patients living with severe obesity receiving Wegovy®.

The TELE-SEMA project involves collecting real-world data on body weight, body composition, cardiovascular and neurovegetative parameters via connected scales in patients with severe obesity treated with Wegovy®.

The main objectives will be to assess inter-individual weight variability and explore the determinants that may influence weight loss, body composition and possible eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged over 18 years
* Patients who have reached the maximum dose of their treatment with Wegovy®
* Written consent

Exclusion Criteria:

* Patient on AME (state medical aid)
* Pregnant or breastfeeding woman
* Patient who does not speak French
* Adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The relative difference in weight loss achieved at 6 months of treatment at the maximum tolerated dose ((weight after 6 months of treatment at the maximum tolerated dose - baseline weight) / baseline weight) | 6 months
  Body weight measured at month 0 and 6

SECONDARY OUTCOMES:
The variation of body weight measured by the connected scale between participants receiving semaglutide at the maximum tolerated dose | 6 months
  Body weight measured weekly
The variation of body composition (fat mass, muscle mass, and bone mass) measured by the connected scale between participants receiving semaglutide at the maximum tolerated dose | 6 months
  Body composition measured weekly
The variation of pulse wave velocity measured by the connected scale between participants receiving semaglutide at the maximum tolerated dose | 6 months
  Pulse wave velocity
The variation of arterial stiffness measured by the connected scale between participants receiving semaglutide at the maximum tolerated dose | 6 months
  Arterial stiffness
The variation of vascular age measured by the connected scale between participants receiving semaglutide at the maximum tolerated dose | 6 months
  Vascular age
The variation of heart rate measured by the connected scale between participants receiving semaglutide at the maximum tolerated dose | 6 months
  Heart rate
The variation of nervous system health (electrochemical skin conductance) measured by the connected scale between participants receiving semaglutide at the maximum tolerated dose | 6 months
  Nervous system health measured weekly
Difference in mean pulse wave velocity before and after 6 months of treatment with semaglutide at the maximum tolerated dose | 6 months
  Pulse wave velocity at month 0 and 6
Difference in mean arterial stiffness before and after 6 months of treatment with semaglutide at the maximum tolerated dose | 6 months
  Arterial stiffness at month 0 and 6
Difference in mean vascular age before and after 6 months of treatment with semaglutide at the maximum tolerated dose | 6 months
  Vascular age at month 0 and 6
Difference in mean heart rate before and after 6 months of treatment with semaglutide at the maximum tolerated dose | 6 months
  Heart rate at month 0 and 6
Difference in eating behavior assessed by the BES questionnaire before and after 6 months of treatment with semaglutide at the maximum tolerated dose | 6 months
  Eating behavior at month 0 and 6
Difference in the level of physical activity assessed by the IPAQ short version questionnaire before and after 6 months of treatment with semaglutide at the maximum tolerated dose | 6 months
  Level of physical activity at month 0 and 6
Percentage of missed doses compared to the total number of prescribed doses after 6 months of treatment at the maximum tolerated dose | 6 months
  missed doses compared to the total number of prescribed doses at month 6

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Czernichow, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital européen Georges Pompidou - APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR)

REFERENCES:
- [Background] World Obesity Federation. World obesity atlas 2022. Ludgate House, London; 2022.
- [Background] ANAES. Rapport sur la chirurgie de l'obésité morbide de l'adulte. 2001.
- [Background] Czernichow S, Renuy A, Rives-Lange C, Carette C, Airagnes G, Wiernik E, Ozguler A, Kab S, Goldberg M, Zins M, Matta J. Evolution of the prevalence of obesity in the adult population in France, 2013-2016: the Constances study. Sci Rep. 2021 Jul 8;11(1):14152. doi: 10.1038/s41598-021-93432-0. PMID 34238998
- [Background] Pan A, Sun Q, Czernichow S, Kivimaki M, Okereke OI, Lucas M, Manson JE, Ascherio A, Hu FB. Bidirectional association between depression and obesity in middle-aged and older women. Int J Obes (Lond). 2012 Apr;36(4):595-602. doi: 10.1038/ijo.2011.111. Epub 2011 Jun 7. PMID 21654630
- [Background] Schneider P, Popkin B, Shekar M, Eberwein JD, Block C, Okamura KS. Health and Economic Impacts of Overweight/Obesity. In: Obesity: Health and Economic Consequences of an Impending Global Challenge [Internet]. The World Bank; 2020 [cited 2021 Nov 5]. p. 69-94. (Human Development Perspectives). Available from: https://elibrary.worldbank.org/doi/10.1596/978-1-4648-1491-4_ch3
- [Background] Thereaux J, Lesuffleur T, Czernichow S, Basdevant A, Msika S, Nocca D, Millat B, Fagot-Campagna A. Long-term adverse events after sleeve gastrectomy or gastric bypass: a 7-year nationwide, observational, population-based, cohort study. Lancet Diabetes Endocrinol. 2019 Oct;7(10):786-795. doi: 10.1016/S2213-8587(19)30191-3. Epub 2019 Aug 2. PMID 31383618
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Wilding JPH, Batterham RL, Calanna S, Van Gaal LF, McGowan BM, Rosenstock J, et al. Impact of Semaglutide on Body Composition in Adults With Overweight or Obesity: Exploratory Analysis of the STEP 1 Study. J Endocr Soc. 2021 May 3;5(Suppl 1):A16-7.
- [Background] Kosiborod MN, Bhatta M, Davies M, Deanfield JE, Garvey WT, Khalid U, Kushner R, Rubino DM, Zeuthen N, Verma S. Semaglutide improves cardiometabolic risk factors in adults with overweight or obesity: STEP 1 and 4 exploratory analyses. Diabetes Obes Metab. 2023 Feb;25(2):468-478. doi: 10.1111/dom.14890. Epub 2022 Oct 28. PMID 36200477
- [Background] Gabery S, Salinas CG, Paulsen SJ, Ahnfelt-Ronne J, Alanentalo T, Baquero AF, Buckley ST, Farkas E, Fekete C, Frederiksen KS, Helms HCC, Jeppesen JF, John LM, Pyke C, Nohr J, Lu TT, Polex-Wolf J, Prevot V, Raun K, Simonsen L, Sun G, Szilvasy-Szabo A, Willenbrock H, Secher A, Knudsen LB, Hogendorf WFJ. Semaglutide lowers body weight in rodents via distributed neural pathways. JCI Insight. 2020 Mar 26;5(6):e133429. doi: 10.1172/jci.insight.133429. PMID 32213703
- [Background] Wharton S, Batterham RL, Bhatta M, Buscemi S, Christensen LN, Frias JP, Jodar E, Kandler K, Rigas G, Wadden TA, Garvey WT. Two-year effect of semaglutide 2.4 mg on control of eating in adults with overweight/obesity: STEP 5. Obesity (Silver Spring). 2023 Mar;31(3):703-715. doi: 10.1002/oby.23673. Epub 2023 Jan 18. PMID 36655300
- [Background] BROWN RE, LIU AR, MAHBUBANI R, ARONSON R. 995-P: Semaglutide in Patients with Type 2 Diabetes: Real-World Analysis in the Canadian LMC Diabetes Registry: The SPARE Study. Diabetes. 2019 Jun 1;68(Supplement_1):995-P.
- [Background] VISARIA J, DANG-TAN T, PETRARO PV, NEPAL BK, WILLEY V. 1006-P: Real-World Effectiveness of Semaglutide in Early Users from a U.S. Commercially Insured (CI) and Medicare Advantage (MA) Population. Diabetes. 2019 Jun 1;68(Supplement_1):1006-P.
- [Background] Di Loreto C, Minarelli V, Nasini G, Norgiolini R, Del Sindaco P. Effectiveness in Real World of Once Weekly Semaglutide in People with Type 2 Diabetes: Glucagon-Like Peptide Receptor Agonist Naive or Switchers from Other Glucagon-Like Peptide Receptor Agonists: Results from a Retrospective Observational Study in Umbria. Diabetes Ther. 2022 Mar;13(3):551-567. doi: 10.1007/s13300-022-01218-y. Epub 2022 Mar 1. PMID 35230650
- [Background] Rajamand Ekberg N, Bodholdt U, Catarig AM, Catrina SB, Grau K, Holmberg CN, Klanger B, Knudsen ST. Real-world use of once-weekly semaglutide in patients with type 2 diabetes: Results from the SURE Denmark/Sweden multicentre, prospective, observational study. Prim Care Diabetes. 2021 Oct;15(5):871-878. doi: 10.1016/j.pcd.2021.06.008. Epub 2021 Jun 25. PMID 34183269
- [Background] Garcia de Lucas MD, Miramontes-Gonzalez JP, Aviles-Bueno B, Jimenez-Millan AI, Rivas-Ruiz F, Perez-Belmonte LM. Real-world use of once-weekly semaglutide in patients with type 2 diabetes at an outpatient clinic in Spain. Front Endocrinol (Lausanne). 2022 Sep 16;13:995646. doi: 10.3389/fendo.2022.995646. eCollection 2022. PMID 36187123
- [Background] Yale JF, Bodholdt U, Catarig AM, Catrina S, Clark A, Ekberg NR, Erhan U, Holmes P, Knudsen ST, Liutkus J, Sathyapalan T, Schultes B, Rudofsky G. Real-world use of once-weekly semaglutide in patients with type 2 diabetes: pooled analysis of data from four SURE studies by baseline characteristic subgroups. BMJ Open Diabetes Res Care. 2022 Apr;10(2):e002619. doi: 10.1136/bmjdrc-2021-002619. PMID 35383100
- [Background] Stewart T, Han H, Allen RH, Bathalon G, Ryan DH, Newton RL Jr, Williamson DA. H.E.A.L.T.H.: efficacy of an internet/population-based behavioral weight management program for the U.S. Army. J Diabetes Sci Technol. 2011 Jan 1;5(1):178-87. doi: 10.1177/193229681100500125. PMID 21303642
- [Background] Beleigoli AM, Andrade AQ, Cancado AG, Paulo MN, Diniz MFH, Ribeiro AL. Web-Based Digital Health Interventions for Weight Loss and Lifestyle Habit Changes in Overweight and Obese Adults: Systematic Review and Meta-Analysis. J Med Internet Res. 2019 Jan 8;21(1):e298. doi: 10.2196/jmir.9609. PMID 30622090
- [Background] Garcia-Ulloa AC, Almeda-Valdes P, Aguilar-Salinas CA, Hernandez-Jimenez S; Group of Study CAIPaDi. Development and Validation of a Software Linked to an Internet Portal That Facilitates the Medical Treatment and Empowerment of Patients with Type 2 Diabetes, Interaction with Medical Personnel, and the Generation of a Real-Time Registry. J Diabetes Sci Technol. 2021 Mar;15(2):525-527. doi: 10.1177/1932296820949941. Epub 2020 Aug 19. No abstract available. PMID 32814459